CLINICAL TRIAL: NCT07349784
Title: Effect of Automated Intraoperative Lung Recruitment Maneuvers on Atelectasis in Patients Undergoing Major Laparoscopic Surgery: A Randomized Controlled Trial
Brief Title: Automated Intraoperative Lung Recruitment Maneuvers in Major Laparoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BakirkoySadiKonukAnesthesia
Record Dates: First submitted 2025-12-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Atelectasis; Postoperative Pulmonary Complications (PPCs)
Keywords: Lung Ultrasound Score (LUS); Automated Lung Recruitment Maneuvers; Laparoscopic Colorectal Surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants assigned to the control group will receive standard intraoperative mechanical ventilation according to institutional practice during general anesthesia for laparoscopic colorectal surgery. No lung recruitment maneuvers will be performed. Perioperative monitoring, anesthetic management, and postoperative care will be standardized and identical to those of the intervention group, except for the application of automated lung recruitment maneuvers.
- Automated Recruitment Group (Experimental): Participants in the intervention group will receive standard intraoperative mechanical ventilation plus automated lung recruitment maneuvers performed by the anesthesia ventilator. The automated recruitment protocol will be applied twice: once after induction of anesthesia and before the initiation of pneumoperitoneum, and once again after pneumoperitoneum is terminated. All other anesthetic management, monitoring, and postoperative care will be identical to the control group.
  Interventions: Procedure: Automated Intraoperative Lung Recruitment Maneuvers

INTERVENTIONS:
Procedure: Automated Intraoperative Lung Recruitment Maneuvers — Automated lung recruitment maneuvers will be performed intraoperatively using the anesthesia ventilator in pressure-controlled ventilation mode according to a standardized protocol.
  Arms: Automated Recruitment Group

SUMMARY:
Laparoscopic colorectal surgery is associated with an increased risk of intraoperative atelectasis due to pneumoperitoneum, Trendelenburg positioning, and prolonged anesthesia duration. Atelectasis developing during surgery may persist into the postoperative period and contribute to postoperative pulmonary complications. Automated lung recruitment maneuvers delivered by modern anesthesia ventilators may offer a standardized method to improve lung aeration and reduce atelectasis. This prospective, randomized, single-center controlled trial aims to evaluate the effect of automated intraoperative lung recruitment maneuvers on atelectasis detected by lung ultrasonography in patients undergoing elective major laparoscopic colorectal cancer surgery. Adult patients will be randomized to receive either automated lung recruitment maneuvers or standard mechanical ventilation without recruitment. Lung ultrasonography will be used to assess atelectasis at predefined perioperative time points. The primary outcome is the incidence of atelectasis detected by lung ultrasound, and secondary outcomes include postoperative pulmonary complications, length of intensive care unit stay, length of hospital stay, and perioperative hemodynamic instability.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-center controlled clinical trial designed to evaluate the effects of automated intraoperative lung recruitment maneuvers on perioperative atelectasis and postoperative pulmonary complications in patients undergoing major laparoscopic colorectal cancer surgery under general anesthesia.

Despite its minimally invasive nature, laparoscopic colorectal surgery is associated with significant perioperative respiratory challenges. Pneumoperitoneum, Trendelenburg positioning, and prolonged operative duration may reduce functional residual capacity, impair respiratory mechanics, and promote intraoperative atelectasis. Atelectasis developing during general anesthesia can persist into the postoperative period and is a major contributor to postoperative pulmonary complications.

Although lung recruitment maneuvers are frequently used to improve lung aeration, manual application lacks standardization and reproducibility. Automated lung recruitment maneuvers delivered by modern anesthesia ventilators may provide a standardized and controlled approach to lung recruitment. Lung ultrasonography is a reliable, bedside, radiation-free imaging modality that allows real-time assessment of lung aeration and detection of atelectasis without the need for patient transport.

After confirmation of eligibility and arrival in the operating room, participants will be randomized in a 1:1 ratio to either an automated lung recruitment maneuver group or a control group receiving standard mechanical ventilation without lung recruitment. Standard intraoperative monitoring will be applied to all patients.

Lung ultrasonography will be used to assess lung aeration and detect atelectasis at predefined perioperative time points, including preoperative baseline assessment, intraoperative evaluation, and postoperative follow-up. Lung ultrasound scores will be used to quantify the degree of aeration loss.

In the intervention group, automated lung recruitment maneuvers will be performed intraoperatively using the anesthesia ventilator according to a standardized protocol. An individualized optimal positive end-expiratory pressure will be determined based on dynamic lung compliance and maintained throughout the surgical procedure. A repeat recruitment maneuver will be applied at the end of surgery after cessation of pneumoperitoneum. The control group will receive standard mechanical ventilation according to institutional practice. Perioperative fluid management will be standardized in both groups using a goal-directed fluid therapy approach.

Postoperative follow-up will include systematic assessment for pulmonary complications. Surgical complications, length of intensive care unit stay, and total hospital length of stay will also be recorded.

The primary outcome of the study is the incidence of atelectasis detected by lung ultrasonography. Secondary outcomes include postoperative pulmonary complications, perioperative hemodynamic instability, length of intensive care unit stay, and length of hospital stay.

This study aims to determine whether automated intraoperative lung recruitment maneuvers assessed using lung ultrasonography can reduce perioperative atelectasis and improve postoperative pulmonary outcomes in patients undergoing major laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Scheduled for elective laparoscopic colorectal cancer surgery
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* ASA physical status IV or higher
* Pregnancy
* Body mass index (BMI) > 40 kg/m²
* Severe chronic obstructive pulmonary disease (COPD), GOLD stage III-IV
* Advanced heart failure with left ventricular ejection fraction <35%
* Previous thoracic surgery
* Preoperative requirement for supplemental oxygen therapy
* Refusal or inability to provide informed consent
* Intraoperative conversion to open surgery
* Development of significant hemodynamic instability during lung recruitment maneuvers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Atelectasis detected by lung ultrasonography | Preoperative baseline (before anesthesia induction), intraoperative assessment (after induction and before pneumoperitoneum), early postoperative assessment (30 minutes after extubation), and postoperative day 1 (within 24 hours after surgery).
  The presence and severity of atelectasis will be assessed using lung ultrasonography performed with a standardized 12-zone scanning protocol. Lung ultrasound scores (LUS) will be calculated for each zone, and severe atelectasis will be defined as a lung ultrasound score of 2 or 3 in any lung region.Lung ultrasound score (LUS) will be assessed using a standardized 12-zone lung ultrasonography protocol. Each lung zone will be scored from 0 to 3 (0 = normal aeration, 1 = moderate loss of aeration, 2 = severe loss of aeration, 3 = consolidation), resulting in a total score ranging from 0 to 36. Higher LUS values indicate worse lung aeration.

SECONDARY OUTCOMES:
Postoperative pulmonary complications | From the end of surgery until hospital discharge (up to postoperative day 30).
  Postoperative pulmonary complications will be defined and classified according to the European Perioperative Clinical Outcome (EPCO) definitions. Complications will include respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonia. Each complication will be diagnosed based on predefined EPCO criteria using clinical findings, imaging studies, laboratory results, and the need for respiratory support or therapeutic interventions.Postoperative pulmonary complications will be assessed daily during hospitalization.
Change in lung ultrasound score (LUS) | From preoperative baseline through postoperative day 1
  Changes in lung ultrasound score will be evaluated using a standardized 12-zone lung ultrasonography protocol. Lung ultrasound scores will be calculated at predefined perioperative time points, and changes in LUS from baseline to intraoperative and postoperative assessments will be analyzed.Lung ultrasound score (LUS) will be assessed using a standardized 12-zone lung ultrasonography protocol. Each lung zone will be scored from 0 to 3 (0 = normal aeration, 1 = moderate loss of aeration, 2 = severe loss of aeration, 3 = consolidation), resulting in a total score ranging from 0 to 36. Higher LUS values indicate worse lung aeration.
Oxygenation parameters (PaO₂/FiO₂ ratio) | Intraoperatively,immediediately after the first recruitment maneuver(within 10 minutes after the maneuver) and during the early postoperative period (30 minutes after extubation).
  Arterial blood gas analyses will be used to assess oxygenation. The PaO₂/FiO₂ ratio will be calculated at predefined perioperative time points to evaluate changes in oxygenation status.

OTHER OUTCOMES:
Length of intensive care unit stay | From postoperative intensive care unit admission until discharge from the intensive care unit (up to 30 days).
  The duration of intensive care unit stay will be recorded in days for patients requiring postoperative intensive care admission.
Length of hospital stay | From the day of surgery until hospital discharge(up to 30 days)
  Total length of hospital stay will be recorded in days from the day of surgery until hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared due to privacy regulations and lack of ethics approval for external data sharing

REFERENCES:
- [Background] Shander A, Fleisher LA, Barie PS, Bigatello LM, Sladen RN, Watson CB. Clinical and economic burden of postoperative pulmonary complications: patient safety summit on definition, risk-reducing interventions, and preventive strategies. Crit Care Med. 2011 Sep;39(9):2163-72. doi: 10.1097/CCM.0b013e31821f0522. PMID 21572323
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Nakahira J, Nakano S, Minami T. Evaluation of alveolar recruitment maneuver on respiratory resistance during general anesthesia: a prospective observational study. BMC Anesthesiol. 2020 Oct 17;20(1):264. doi: 10.1186/s12871-020-01182-9. PMID 33069208
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555
- [Background] Yu X, Zhai Z, Zhao Y, Zhu Z, Tong J, Yan J, Ouyang W. Performance of Lung Ultrasound in Detecting Peri-Operative Atelectasis after General Anesthesia. Ultrasound Med Biol. 2016 Dec;42(12):2775-2784. doi: 10.1016/j.ultrasmedbio.2016.06.010. Epub 2016 Sep 14. PMID 27639431